CLINICAL TRIAL: NCT05280353
Title: Seroma Control in Axillary Lymphadenectomy With Glubran 2® Without Drain. Multicenter, Prospective, Randomized Clinical Trial. GALA-ND Study (Glu Axillary Lymphadenectomy Ambulatory- no Drain)
Brief Title: Use of Glubran 2 ® in Axillary Lymphadenectomy Without Drain
Acronym: GALA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Omphis Foundation (Other)
Collaborators: Consorci Sanitari del Maresme (Other)
Responsible Party: Principal Investigator, Sandra Lopez Gordo, Principal investigator, Omphis Foundation
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Health consortium maresme
Record Dates: First submitted 2022-02-08; First posted 2022-03-15 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Seroma Following Procedure
MeSH Terms: interventions — glubran 2

STUDY DESIGN:
Intervention Model Description: MULTICENTRIC, PROSPECTIVE, RANDOMIZED CLINICAL TRIAL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lymphadenectomy without drainage and with Glubran (Experimental): Application of Glubran 2 in axillary dissection with the objective of seroma reduction. No drain
  Interventions: Other: Glubran 2
- Lymphadenectomy without drainage (No Intervention): No intervention required, only axillary dissection without drain

INTERVENTIONS:
Other: Glubran 2 — Application of Glubran 2 sealant (liquid) in axillary hollow
  Arms: lymphadenectomy without drainage and with Glubran

SUMMARY:
Axillary lymphadenectomy in breast cancer continues to be a common practice in certain patients. The use of sealants and drains continues to be a source of disagreement among the scientific community. That is why the study was designed to show whether the sealant reduces seroma after axillary lymphadenectomy without drainage.

DETAILED DESCRIPTION:
A study has been designed to assess whether the sealant reduces the rate of symptomatic seroma measured by the number of evacuating punctures. Likewise, the decrease in volume due to the seroma between the two groups and the quality of life of the patients is assessed, given that none of them has a drain

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Conservative surgery for breast cancer with associated axillary lymphadenectomy

Exclusion Criteria:

* Mastectomy
* History of axillary surgery or ipsilateral axillary radiotherapy
* ASA 4 patients. (ASA 3 patients selected)
* Lack of adequate cognitive capacity and/or signed informed consent
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in symptomatic seroma | Up tp 1 year
  Number of evacuating punctures
Number of participants with treatment-related adverse events | Up to 1 year
  Type and number of adverse events

SECONDARY OUTCOMES:
Seroma volume | Day 7 and 14 after surgery
  Volume measured by ultrasound (cm3 )
Milliliters of evacuated seroma in case of puncture | 7, 14 and 30 day after surgery
  Assess if there are differences in the volume of seroma evacuated (milliliters) between groups
Demographic characteristics of patients related to seroma | Up to 1 year
  Assess the existence of risk factors (age, sex, obesity,neoadjuvant treatment) related to symptomatic seroma
Number of patients with temporary or permanence of disability after operation | Up to 1 year
  Clavien-Dindo classification of morbidity
Individual's perception of the position in life of the participants | Day 7 and 14 after surgery
  Assess the quality of life after the intervention measured by the EuroQol five dimensions (EQ-5D-5L questionnaire). Descriptive system for health-related quality of life states in adults, consisting of five dimensions. No quality 0 points. Perfect quality 100 points

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lopez Gordo, Doctor, Principal Investigator — Health Consortium Maresme
Locations (1):
- Maresme health consortium, Mataró, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giuliano AE, Ballman KV, McCall L, Beitsch PD, Brennan MB, Kelemen PR, Ollila DW, Hansen NM, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, Hunt KK, Morrow M. Effect of Axillary Dissection vs No Axillary Dissection on 10-Year Overall Survival Among Women With Invasive Breast Cancer and Sentinel Node Metastasis: The ACOSOG Z0011 (Alliance) Randomized Clinical Trial. JAMA. 2017 Sep 12;318(10):918-926. doi: 10.1001/jama.2017.11470. PMID 28898379
- [Background] van Bemmel AJ, van de Velde CJ, Schmitz RF, Liefers GJ. Prevention of seroma formation after axillary dissection in breast cancer: a systematic review. Eur J Surg Oncol. 2011 Oct;37(10):829-35. doi: 10.1016/j.ejso.2011.04.012. Epub 2011 Aug 17. PMID 21849243
- [Background] Srivastava V, Basu S, Shukla VK. Seroma formation after breast cancer surgery: what we have learned in the last two decades. J Breast Cancer. 2012 Dec;15(4):373-80. doi: 10.4048/jbc.2012.15.4.373. Epub 2012 Dec 31. PMID 23346164
- [Background] Thomson DR, Sadideen H, Furniss D. Wound drainage after axillary dissection for carcinoma of the breast. Cochrane Database Syst Rev. 2013 Oct 20;2013(10):CD006823. doi: 10.1002/14651858.CD006823.pub2. PMID 24158902
- [Background] Chang YT, Shih SL, Loh EW, Tam KW. Effects of Fibrin Sealant on Seroma Reduction for Patients with Breast Cancer Undergoing Axillary Dissection: Meta-Analysis of Randomized Controlled Trials. Ann Surg Oncol. 2020 Dec;27(13):5286-5295. doi: 10.1245/s10434-020-08747-5. Epub 2020 Jun 20. PMID 32564232
- [Background] Gunn J, Gibson T, Li Z, Diehl N, Bagaria S, McLaughlin S. Symptomatic Axillary Seroma after Sentinel Lymph Node Biopsy: Incidence and Treatment. Ann Surg Oncol. 2016 Oct;23(10):3347-53. doi: 10.1245/s10434-016-5398-6. Epub 2016 Jul 8. PMID 27393569
- [Background] Jain PK, Sowdi R, Anderson AD, MacFie J. Randomized clinical trial investigating the use of drains and fibrin sealant following surgery for breast cancer. Br J Surg. 2004 Jan;91(1):54-60. doi: 10.1002/bjs.4435. PMID 14716794
- [Background] Vasileiadou K, Kosmidis C, Anthimidis G, Miliaras S, Kostopoulos I, Fahantidis E. Cyanoacrylate Adhesive Reduces Seroma Production After Modified Radical Mastectomy or Quadrantectomy With Lymph Node Dissection-A Prospective Randomized Clinical Trial. Clin Breast Cancer. 2017 Dec;17(8):595-600. doi: 10.1016/j.clbc.2017.04.004. Epub 2017 Apr 13. PMID 28673765
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. J Clin Epidemiol. 2009 May;62(5):464-75. doi: 10.1016/j.jclinepi.2008.12.011. PMID 19348971
- [Derived] Lopez Gordo S, Ruiz-Edo N, Fernandez-Planas MT, Viscaya-Martin S, Serra-Serra C; Breast Cancer Research Group. Seroma control in axillary lymphadenectomy with Glubran 2(R) without drain. Multicenter, prospective, randomized, clinical trial. GALA-ND study (Glubran, Axillary Lymphadenectomy, Ambulatory, No Drain). Trials. 2024 Feb 22;25(1):142. doi: 10.1186/s13063-023-07840-w. PMID 38388444